CLINICAL TRIAL: NCT03036930
Title: Immunogenicity of Nonavalent HPV Vaccine Administered Prior to Renal Transplantation in Adults: A Prospective, Single-Arm, Multi-Center Clinical Trial
Brief Title: Preventive Human Papillomavirus (HPV) Vaccine Trial in Kidney Transplant Recipients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2017-00116; NCI-2017-00116 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00035; NCI2015-06-02 (Other: Northwestern University); NWU2015-06-02 (Other: DCP); N01CN00035 (NIH); P30CA060553 (NIH)
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Results first posted 2025-12-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Human Papillomavirus Infection; Human Papillomavirus-Related Carcinoma
MeSH Terms: conditions — Papillomavirus Infections | interventions — Specimen Handling; Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (Gardasil 9 HPV vaccine) (Experimental): Participants receive the first dose of the recombinant human papillomavirus nonavalent vaccine IM at baseline, at least 30 days prior to the kidney transplant surgery. The second dose is given at least one month after the first dose. The third dose is given at least five months after the first dose and at least three months after the second dose. The timing of the second and third doses is dependent on the scheduling of the kidney transplant surgery. Patients are followed up at 6- and 12-months after the kidney transplant surgery to measure vaccine-induced immune responses. Patients may receive either one, two, or all three vaccine doses prior to the kidney transplant surgery, and are offered additional visits at least one year after the surgery to complete any remaining doses of the three-dose vaccine series. Patients also undergo collection of blood samples and self-collection of cervical/vaginal samples (female participants only) on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: HPV Self-Collection; Other: Questionnaire Administration; Biological: Recombinant Human Papillomavirus Nonavalent Vaccine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: HPV Self-Collection — Undergo self-collection of vaginal/cervical samples
  Other Names: At-home HPV Self Collection; HPV Self Collection; Human Papillomavirus Self-Collection
Other: Questionnaire Administration — Ancillary studies
Biological: Recombinant Human Papillomavirus Nonavalent Vaccine — Given IM
  Other Names: Gardasil 9; Nonavalent HPV VLP Vaccine; Recombinant HPV Nonavalent Vaccine; Recombinant Human Papillomavirus 9-valent Vaccine

SUMMARY:
This phase II trial studies whether the nonavalent human papillomavirus vaccine given to adults prior to kidney transplantation can help the body build and maintain an effective immune response during the post-transplant period when they receive immunosuppressive drugs to prevent transplant rejection. This study will help inform our scientific understanding about vaccine-induced immune responses among immunosuppressed individuals.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess human papillomavirus (HPV) vaccine-type-specific seroconversion rates at 12-months post-transplantation among kidney transplant recipients who receive >= 1 doses of the recombinant human papillomavirus nonavalent vaccine (Gardasil [registered trademark] 9 HPV vaccine) >= 30 days prior to transplantation.

SECONDARY OBJECTIVE:

I. To assess HPV vaccine-type-specific seroconversion rates at 6- and 12-months post-transplantation stratified by number of doses (1, 2, or 3) of the vaccine given pre-transplant among kidney transplant recipients who receive >= 1 doses of the Gardasil 9 HPV vaccine prior to transplantation.

EXPLORATORY OBJECTIVES:

I. To assess the following among kidney transplant recipients who receive >= 1 doses of the Gardasil 9 HPV vaccine >= 30 days prior to transplantation:

Ia. HPV vaccine-type-specific seroconversion rates at 12-months post-transplantation stratified by:

Ii. Time elapsed between last vaccine dose and the transplant procedure; Iii. Variations in dosing and types of post-transplant immunosuppressant medications; and interactions with type of transplant surgery (living donor/deceased donor); Iiii. Differences in human leukocyte antigen (HLA) histocompatibility between donor and recipient; Iiv. Differences in biological sex (i.e. male versus [vs.] female) of the transplant recipient; Ib. Stability of HPV vaccine-type-specific geometric mean titers (GMT) at 6 and 12-months post-transplantation and rise in HPV vaccine-type-specific GMT at the 13-month post-transplant visit; Ic. Vaccine safety profile and allograft rejection/opportunistic infections stratified by number of vaccine doses and time between the last vaccine dose and the transplant procedure; Id. HPV detection in samples from the cervix/vagina and oral cavity at baseline (pre-vaccination) and at 6- and 12-months post-vaccination, overall and by number of vaccine doses (1, 2, or 3), sexual behavior, type-specific seroconversion rates, and time elapsed between the last vaccine dose and the transplant procedure.

OUTLINE:

Participants receive the first dose of the recombinant human papillomavirus nonavalent vaccine intramuscularly (IM) at baseline, at least 30 days prior to the kidney transplant surgery. The second dose is given at least one month after the first dose. The third dose is given at least five months after the first dose and at least three months after the second dose. The timing of the second and third doses is dependent on the scheduling of the kidney transplant surgery. Patients are followed up at 6- and 12-months after the kidney transplant surgery to measure vaccine-induced immune responses. Patients may receive either one, two, or all three vaccine doses prior to the kidney transplant surgery, and are offered additional visits at least one year after the surgery to complete any remaining doses of the three-dose vaccine series. Patients also undergo collection of blood samples and self-collection of cervical/vaginal samples (female participants only) on study.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for renal transplant, expected to undergo transplant surgery >= 30 days and =< 12 months after enrollment

  * For potential participants on the institutional waiting list for deceased donor transplant, a study clinician confirms the candidate is likely to receive a transplant within the next 12 months, taking into account the candidate's priority on the waiting list, age, medical status, institutional policies, and scores like the Estimated Post-Transplant Survival (EPTS) Score and Calculated Panel Reactive Antibody (CPRA) percentage, etc
  * For potential participants expected to undergo a living donor transplant, one or more donor(s) have been identified and is/are in work-up (even though all work-up status may or may not be complete); a study clinician confirms the living donor transplant is likely to be scheduled within the next twelve months after taking into account donor work-up progress, age and medical status, and institutional policies
  * Notes:

    * Living and deceased donor transplant recipients: The study was originally restricted to participants who were expecting to receive only living donor renal transplants; however, less than a third of kidney transplants in the United States occur with kidneys from living donors; a majority of transplants are in the setting of donation of kidneys from deceased donors; to permit efficiencies in accrual, the study is amended (from version 3.5) to also open enrollment to recipients of deceased donor kidneys
    * Transplant recipients of both genders: The study was originally designed to be conducted only among women; however, in October 2018, the Food and Drug Administration (FDA) approved an age expansion indication for the Gardasil 9 HPV vaccine for both women and men up to 45 years (from the originally approved upper age limit of 26 years), thus opening a new clinical cancer preventative option for middle-age adults of both genders; the primary endpoint for the study is HPV-vaccine-type-specific seroconversion rates, which are not expected to be differential by gender, based on extrapolating from the uniformly high (> 99%) seroconversion rates observed regardless of gender in studies among immunocompetent individuals; however, HPV vaccine-type-specific titer levels (GMT) differences by gender will be analyzed as a secondary endpoint, given variability in immune response titer levels observed between males and females in immunocompetent individuals (related to the differences in body mass index or hitherto unproven factors related to hormone-immune interactions); another advantage of expanding this study to males will be to facilitate efficiencies in accrual, since men constitute the majority (55%-65%) of all kidney transplant recipients in the United States; although a majority of current HPV-associated cancers among solid organ transplant recipients occur among women, there is increasing evidence of the link between HPV infection and oropharyngeal cancers that disproportionately affect men; HPV-related oropharyngeal cancers are now the most common HPV-related cancers in the United States, surpassing even the incidence of cervical cancer; the expansion of enrollment to men will also allow this study to look at the effect of HPV vaccination on persistence of oral HPV infection as a secondary/exploratory endpoint in the context of transplant-related immunosuppression
* Age 18-49 years. We have chosen to focus on adults aged 18-49 for this initial study in transplant recipients for a few reasons. Prior data for HPV vaccine response exists for adults up to 49 years of age, providing an important external comparison group for our study. Immune response and exposure wane as age increases and we want to minimize the potential for age-related confounding of our study outcome. For this initial trial, we thought it best to maintain homogeneity in the study population to the extent possible. Finally, given that about half of renal transplant recipients in the United States (U.S.) are between the ages of 18-49 years, selecting this age range permits efficiency in study accrual
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* The effects of the Gardasil 9 HPV vaccine on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because there have been no adequate and well-controlled studies of Gardasil 9 in pregnant women, women who are able to become pregnant must have a confirmed negative pregnancy test result within the past 28 days prior to enrollment and must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; women who have had a both ovaries removed or a tubal ligation will not be required to have a pregnancy test; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document and medical release form
* Willing and able to comply with trial protocol and follow-up

Exclusion Criteria:

* Previous prophylactic HPV vaccination
* Prior organ transplant
* Anticipated desensitization treatment; this decision to exclude a participant who may need desensitization will be based on the site clinician's judgement; desensitization procedures vary somewhat among the five participating transplant centers, which does not permit proposing uniform criteria across all study sites for determining exclusion due to desensitization; in general, women who have received a prior transplant, have unsuitable scores on Calculated Panel Reactive Antibody (PRA) percentage (institution-specific thresholds), or an ABO incompatible donor are likely to undergo desensitization at one or more of the study centers; these factors, among others, will be used by the study clinician to determine exclusion due to anticipated desensitization is warranted for a particular participant in the study
* Current use of any other investigational agents
* History of allergic reactions to yeast or attributed to compounds of similar chemical or biologic composition to Gardasil 9 HPV vaccine
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* For female participants: Pregnant or intention to get pregnant, or breastfeeding; pregnant women are excluded from this study because the safety and effectiveness of Gardasil 9 HPV vaccine have not been established in pregnant women; it is not known whether Gardasil 9 is excreted in human milk; because many drugs are excreted in human milk, caution should be exercised when Gardasil 9 is administered to a nursing woman; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Gardasil 9, women who are breastfeeding will be excluded
* History of cervical cancer or anal cancer
* History of active malignancy, including basal/squamous cell skin cancer
* Concurrent illness, such as known psychiatric disorders or substance abuse (i.e., average alcohol consumption of more than 3 drinks per day), which in the opinion of the investigators would compromise either the patient or the integrity of the data
* Patients on anticoagulation or with bleeding disorders should be evaluated by a physician for risk/benefit of bleeding disorders with intramuscular injections prior to study enrollment; patients determined to be at high risk for bleeding with intramuscular injections will be excluded

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2026-03-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marc T Goodman, Principal Investigator — Northwestern University
Locations (6):
- United States (6):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevention (Gardasil 9 HPV Vaccine)
Started | 51
Completed | 26
Not Completed | 25
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 3
Not completed — Not eligible to receive transplant within 12 months | 15

BASELINE CHARACTERISTICS:
Population: Eligible participants registered and enrolled to the trial.
Arm/Group | Prevention (Gardasil 9 HPV Vaccine)
Number analyzed (Participants) | 51
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [33 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 26
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51
Number of Gardasil 9 Doses Before Kidney Transplant [Count of Participants; unit: Participants]
  One | 5
  Two | 14
  Three | 13
  No Transplant | 19

OUTCOME MEASURES:

1. Primary Outcome: HPV Vaccine-type-specific Seroconversion Rates Among Kidney Transplant Recipients Who Received ≥ 1 Doses of the Vaccine.
Description: An estimate of the Human papillomavirus (HPV) vaccine-type-specific seroconversion rate provided along with exact Clopper-Pearson 95% confidence intervals (CIs). All participants who received a kidney transplant were included in the primary endpoint analysis, regardless of whether the last vaccine dose was administered ≥ 30 days prior to transplantation.
Time Frame: At 12 months post-transplant
Population: Participants with HPV labs available 12 months post-transplant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prevention (Gardasil 9 HPV Vaccine)
Number analyzed (Participants) | 20
percentage of participants
  HPV 6 | 70 [45.7 to 88.1]
  HPV 11 | 95 [75.1 to 99.9]
  HPV 16 | 90 [68.3 to 98.8]
  HPV 18 | 65 [40.8 to 84.6]
  HPV 31 | 90 [68.3 to 98.8]
  HPV 33 | 90 [68.3 to 98.8]
  HPV 45 | 50 [27.2 to 72.8]
  HPV 52 | 45 [23.1 to 68.5]
  HPV 58 | 85 [62.1 to 96.8]
  HPV All 9 Subtypes | 25 [8.7 to 49.1]
  HPV ≥ 1 Subtype | 95 [75.1 to 99.9]

2. Secondary Outcome: To Assess HPV Vaccine-type-specific Seroconversion Rates at 6-months Post-transplantation Stratified by Number of Doses (1, 2, or 3) Given Pre-transplant Among Kidney Transplant.
Description: An estimate of the HPV vaccine-type-specific seroconversion rates at 6-months post-transplantation stratified by number of doses (1, 2, or 3) of the vaccine given pre-transplant was provided along with 95% confidence intervals (CIs). Clopper-Pearson CIs were provided for the overall and stratified estimates.
Time Frame: At 6-months post-transplant
Population: Participants with HPV labs available 6 months post-transplant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- One Pre-Transplant Dose: Kidney transplant recipients who received 1 dose of the HPV vaccine ≥ 30 days prior to transplantation.
- Two Pre-Transplant Doses: Kidney transplant recipients who received 2 doses of the HPV vaccine ≥ 30 days prior to transplantation.
- Three Pre-Transplant Doses: Kidney transplant recipients who received 3 doses of the HPV vaccine ≥ 30 days prior to transplantation.
- Overall Pre-Transplants Doses: Kidney transplant recipients who receive ≥ 1 doses of the HPV vaccine ≥ 30 days prior to transplantation.
Arm/Group | One Pre-Transplant Dose | Two Pre-Transplant Doses | Three Pre-Transplant Doses | Overall Pre-Transplants Doses
Number analyzed (Participants) | 3 | 10 | 10 | 23
percentage of participants
  HPV 6 | 100 [43.9 to 100] | 30 [10.8 to 60.3] | 90 [59.6 to 98.2] | 65.2 [42.7 to 83.6]
  HPV 11 | 100 [43.9 to 100] | 70 [39.2 to 89.2] | 100 [72.2 to 100] | 87 [66.4 to 97.2]
  HPV 16 | 100 [43.9 to 100] | 90 [59.6 to 98.2] | 100 [72.2 to 100] | 95.7 [78.1 to 99.9]
  HPV 18 | 66.7 [20.8 to 93.9] | 70 [39.7 to 89.2] | 80 [49 to 94.3] | 73.9 [51.6 to 89.9]
  HPV 31 | 66.7 [20.8 to 93.9] | 80 [49 to 94.3] | 90 [59.6 to 98.2] | 82.6 [61.2 to 95]
  HPV 33 | 66.7 [20.8 to 93.9] | 90 [59.6 to 98.2] | 90 [59.6 to 98.2] | 87 [66.4 to 97.2]
  HPV 45 | 66.7 [20.8 to 93.9] | 20 [5.7 to 51] | 90 [59.6 to 98.2] | 56.5 [34.5 to 76.8]
  HPV 52 | 66.7 [20.8 to 93.9] | 30 [10.8 to 60.3] | 60 [31.3 to 83.2] | 47.8 [26.8 to 69.4]
  HPV 58 | 66.7 [20.8 to 93.9] | 70 [39.7 to 89.2] | 80 [49 to 94.3] | 73.9 [51.6 to 89.8]
  HPV All 9 Subtypes | 66.7 [20.8 to 93.9] | 10 [1.8 to 40.4] | 50 [23.7 to 76.3] | 34.8 [16.4 to 57.3]
  HPV ≥ 1 Subtype | 100 [43.9 to 100] | 90 [59.6 to 98.2] | 100 [72.2 to 100] | 95.7 [78.1 to 99.9]

3. Other Pre Specified Outcome: Probability of Seroconversion
Description: Descriptive statistics, such as probabilities and exact 95% CIs, will be used to summarize probability of seroconversion at 12 months post-transplant for the following groups: a) time elapsed between last vaccine dose and the transplant procedure, e.g. < 3 months versus (vs.) > 3 months. Different groupings will be considered based on observed (e.g. median) and clinical considerations. Time will be summarized using descriptive statistics, e.g. median, interquartile range, or range; groups defined by dosing and types of post-transplant immunosuppressant medications, as well as; b) type of transplant surgery (living donor/deceased donor); c) differences in human leukocyte antigen histocompatibility between donor and recipient; d) differences by biological sex (i.e., male vs. female) of the transplant recipient.
Time Frame: At 12 months post-transplant
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Stability of HPV Vaccine-type-specific Geometric Mean Titers (GMT)
Description: Stability will be evaluated in relation to changes in the type-specific GMTs between the two post-transplant time points (6- and 12-months post-transplant) and reported as follows: (i) decrease: more than 2-fold decrease, (ii) stable: within 2-fold change, and (iii) increase: greater than 2-fold increase. Stability will also be described in relation to the number of vaccine doses (1, 2 or 3) received in the pre-transplant period.
Time Frame: At 6 and 12 months post-transplant
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Rise in HPV Vaccine-type-specific GMT
Description: The magnitude of increase in type-specific GMTs at the 13-month post-transplant visit (i.e., 1 month after the booster dose) will be described in relation to the type-specific GMTs at the other post-transplant visits (6 and 12-months post -transplant). Patterns over time will also be explored using graphical techniques. Post-booster dose increase in type-specific GMTs will also be described in relation to the number of vaccine doses (1, 2 or 3) received in the pre-transplant period.
Time Frame: At 13 months post-transplant
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Vaccine Safety Profile and Allograft Rejection/Opportunistic Infections
Description: Will be summarized using descriptive statistics, stratified by number of vaccine doses and time between the last vaccine dose and the transplant procedure.
Time Frame: Up to 13 months post-transplant
Reporting Status: Not Posted

7. Other Pre Specified Outcome: HPV Detection in Samples From the Cervix/Vagina, and Oral Cavity
Description: HPV detection in samples from the cervix/vagina, and oral cavity at baseline (pre-vaccination) and at 6- and 12-months post-vaccination, overall and by number of vaccine doses (1, 2, or 3), sexual behavior, type-specific seroconversion rates, and time elapsed between the last vaccine dose and the transplant procedure will be evaluated. All rates of HPV detection will be specified, overall and stratified by number of doses (1, 2, or 3) and time to transplant.
Time Frame: Self-collected at baseline (pre-vaccination) and at 6- and 12- months post-vaccination
Reporting Status: Not Posted

8. Secondary Outcome: To Assess HPV Vaccine-type-specific Seroconversion Rates at 12-months Post-transplantation Stratified by Number of Doses (1, 2, or 3) Given Pre-transplant Among Kidney Transplant.
Description: An estimate of the HPV vaccine-type-specific seroconversion rates at 12-months post-transplantation stratified by number of doses (1, 2, or 3) of the vaccine given pre-transplant was provided along with 95% confidence intervals (CIs). Clopper-Pearson CIs were provided for the overall and stratified estimates.
Time Frame: At 12- months post-transplant
Population: Participants with HPV labs available 12 months post-transplant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | One Pre-Transplant Dose | Two Pre-Transplant Doses | Three Pre-Transplant Doses | Overall Pre-Transplants Doses
Number analyzed (Participants) | 2 | 9 | 9 | 20
percentage of participants
  HPV 6 | 100 [15.8 to 100] | 55.6 [21.2 to 86.3] | 77.8 [40 to 97.2] | 70 [45.7 to 88.1]
  HPV 11 | 100 [15.8 to 100] | 88.9 [51.8 to 99.7] | 100 [66.4 to 100] | 95 [75.1 to 99.9]
  HPV 16 | 100 [15.8 to 100] | 88.9 [51.8 to 99.7] | 88.9 [51.8 to 99.7] | 90 [68.3 to 98.8]
  HPV 18 | 100 [15.8 to 100] | 44.4 [13.7 to 78.8] | 77.8 [40 to 97.2] | 65 [40.8 to 84.6]
  HPV 31 | 100 [15.8 to 100] | 88.9 [51.8 to 99.7] | 88.9 [51.8 to 99.7] | 90 [68.3 to 98.8]
  HPV 33 | 100 [15.8 to 100] | 88.9 [51.8 to 99.7] | 88.9 [51.8 to 99.7] | 90 [68.3 to 98.8]
  HPV 45 | 100 [15.8 to 100] | 33.3 [7.5 to 70.1] | 55.6 [21.2 to 86.3] | 50 [27.2 to 72.8]
  HPV 52 | 100 [34.2 to 100] | 55.6 [21.2 to 86.3] | 22.2 [2.8 to 60] | 45 [23.1 to 68.5]
  HPV 58 | 100 [15.8 to 100] | 88.9 [51.8 to 99.7] | 77.8 [40 to 97.2] | 85 [62.1 to 96.8]
  HPV All 9 Subtypes | 100 [15.8 to 100] | 22.2 [2.8 to 60] | 11.1 [0.3 to 48.2] | 25 [8.7 to 49.1]
  HPV ≥ 1 Subtype | 100 [15.8 to 100] | 88.9 [51.8 to 99.7] | 100 [66.4 to 100] | 95 [75.1 to 99.9]

ADVERSE EVENTS:
Time Frame: Pre-transplant up to 15 months post-transplant.
Groups:
- Prevention (Gardasil 9 HPV Vaccine): Participants receive the first dose of the recombinant human papillomavirus nonavalent vaccine IM at baseline, at least 30 days prior to the kidney transplant surgery. The second dose is given at least one month after the first dose. The third dose is given at least five months after the first dose and at least three months after the second dose. The timing of the second and third doses is dependent on the scheduling of the kidney transplant surgery. Participants are followed up at 6- and 12-months after the kidney transplant surgery to measure vaccine-induced immune responses. Participants may receive either one, two, or all three vaccine doses prior to the kidney transplant surgery, and are offered additional visits at least one year after the surgery to complete any remaining doses of the three-dose vaccine series. Participants also undergo collection of blood samples and self-collection of cervical/vaginal samples (female participants only) on study.
  Biospecimen Collection: Undergo collection of blood samples
  HPV Self-Collection: Undergo self-collection of vaginal/cervical samples
  Questionnaire Administration: Ancillary studies
  Recombinant Human Papillomavirus Nonavalent Vaccine: Given IM
Arm/Group | Prevention (Gardasil 9 HPV Vaccine)
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 8/51
Other Adverse Events (participants affected / at risk) | 26/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevention (Gardasil 9 HPV Vaccine) (N=51)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — New onset diabetes mellitus
Sepsis (Infections and infestations) | 1 (1) — Culture negative sepsis
Abdominal infection (Infections and infestations) | 1 (1) — Tunnel infection
Hypertension (Vascular disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) — Congestive heard failure
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — COVID-19 documented with fever
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevention (Gardasil 9 HPV Vaccine) (N=51)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Headache (Nervous system disorders) | 6 (6)
Infections and infestations - Other, specify (Infections and infestations) | 6 (6) — COVID-19 (4)
Injection site reaction (General disorders) | 11 (12)
Nausea (Gastrointestinal disorders) | 4 (4)
Paresthesia (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT03036930/Prot_SAP_ICF_001.pdf